CLINICAL TRIAL: NCT03628859
Title: BIOREN (Predictive BIOmarkers in Metastatic RENal Cancer) - A Translational Study on Immunotherapy for Metastatic Renal Cancer
Brief Title: BIOREN (Predictive BIOmarkers in Metastatic RENal Cancer)
Acronym: BIOREN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: BIOREN (ET18-017)
Record Dates: First submitted 2018-03-28; First posted 2018-08-14 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Renal Cancer Metastatic
Keywords: Renal cancer metastatic; Immunotherapy; Predictive biomarkers; Translational study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Archival FFPE specimen
  Blood samples performed during standard visits and not requiring additional blood tests:
  * Heparin blood (4 x 6ml)
  * EDTA blood (5 x 6ml)
  * Liquid biopsy (EDTA) (5 x 6ml)
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Immunological and tumour characterization — FFPE, blood samples (liquid biopsy, heparin and EDTA blood) performed in patients presenting a renal metastatic cancer receiving treatment as standard practice according to physician's choice (2nd or 3rd line of treatment with nivolumab, everolimus, axitinib or cabozantinib [in France only], as per product SmPC or 1st line treatment with sunitinib or pazopanib or receiving 2nd or 3rd line of treatment with nivolumab)

SUMMARY:
The BIOREN project aims are to characterize the genetic background of renal cell carcinomas and their immune environment, to try and identify biomarkers of response and to better understand the mechanisms of resistance to nivolumab in renal cancer.

DETAILED DESCRIPTION:
Around 338,000 new cases of renal cell carcinoma (RCC) are diagnosed worldwide per year (1). RCC is one of the most immune responsive human cancers. For a long time the only available treatment were high-dose IL-2 and IFN-α with only a few patients achieving durable responses. Clinical trials conducted in the past 15 years have led to the approval of several anti-angiogenic treatments, mainly vascular endothelial growth factor receptor (VEGFR) inhibitors and mTOR inhibitors. Currently most patients receive first line anti-VEGF therapy.

Recently a better understanding of the mechanisms by which tumours evade the immune system has led to the development of checkpoint inhibitors, such as anti CTLA-4, anti-PD-1 and anti-PD-L1 antibodies that have been tested in various tumour types.

Recently, the US Food and Drug Administration (FDA) and the European Medicines Agency (EMA) have approved the human IgG4 anti-PD1 monoclonal antibody, nivolumab, for advanced/metastatic clear cell RCC (ccRCC) patients who have received prior antiangiogenic therapy. PD-1 is a key immune-checkpoint receptor (ICR) expressed by activated T cells, which mediates immunosuppression primarily in peripheral tissues, where T cells may encounter the immunosuppressive PD-1 ligands, PD-L1 (B7-H1) and PD-L2(B7-DC) on tumour cells, stromal cells or both.

Despite encouraging results, the clinical response to anti-PD1 is not as wide as expected and there are not any biomarkers 1) that are able to predict which patients will respond and 2) that predict response to nivolumab in patients with ccRCC.

BIOREN is a translational, prospective, observational 3-cohort study.

The aims of BIOREN are to characterize the genetic background of the tumours and also their immune environment, to try and identify biomarkers of response and to better understand the mechanisms of resistance to nivolumab in renal cancer. We will focus on:

* Tregs function and modulation of function,
* NK cells known to be regulated by nivolumab,
* The biological rationale for coupling CXCR4 antagonist with anti PD-1 therapy, analysed with mice models,
* To try to identify biomarkers of response by further characterization of the tumours and evaluating the immune status.

The project will enrol patients receiving in 2nd or 3rd line treatment for metastatic ccRCC: Nivolumab but also, as control cohorts, either everolimus or axitinib (approved treatments in this setting), as well as cabozantinib in France (recently approved in 2nd or 3rd line).

French blood samples and archival FFPE (formalin-fixed paraffin embedded) specimens will be analysed in in France, and also sent to the partners of the Transcan project Consortium (Israel, Italy and Spain).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years-old.
* Histology proven locally advanced (unresectable) or metastatic clear cell renal cell carcinoma (mccRCC).
* Starting 2nd or 3rd line of treatment with nivolumab, everolimus, axitinib or cabozantinib as per summaries of product characteristics (SmPC) or 1st line treatment with sunitinib or pazopanib or receiving 2nd or 3rd line of treatment with nivolumab
* Signed informed consent.

Exclusion Criteria:

* Psychological, familial, sociological, geographical conditions that would limit compliance with study protocol requirements.
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting a renal metastatic cancer included in Centre Leon Berard for evaluating the mechanisms involved in resistance to immunotherapy:
  * Cohort 1: ccRCC patients receiving nivolumab,
  * Cohort 2: ccRCC patients receiving axitinib or cabozantinib or sunitinib or pazopanib,
  * Cohort 3: ccRCC patients receiving everolimus.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Tregs function on peripheral blood/neoplastic tissue from mRCC patients undergoing nivolumab treatment | Evolution of percentage of CD4+CD25+ CD127low FOXP3+ cells between inclusion and up to 24 months
  Ex vivo effect of CXCR4 antagonists (PCT/IB2011/000120/ EP2528936B1/ US2013/0079292A1) and other Tregs targets antagonists (ICOS, CD39/CD73) or agonists (TLR7L) as putative anti-PD1 resistance mechanisms

SECONDARY OUTCOMES:
Evaluation of NK function/cytotoxicity on peripheral blood/neoplastic tissue from mRCC patients undergoing nivolumab treatment | Evolution between inclusion and up to 24 months
  NK cytotoxicity will be evaluated through NK cell degranulation (CD107a assay), intracellular staining of the lytic proteins, Grz A and GrzB and intracellular cytokines, GM-CSF, IFNγ, IL-10, TNF. NK cell will be characterized for CXCR4; maturation markers: CD16, CD56, CD57, CD62L, NKG2A; activating receptors markers: CD25, CD69, NKp44, NKp30, NKp46, NKG2D. Ex vivo effect of CXCR4 antagonists on NK cytotoxicity.
Exploration of the biological rationale for coupling CXCR4 antagonist with anti-PD-1 in in vivo models of renal cancer (mice models). | Up to 24 months
  immunocompetent model (RENCA), human xenograft model (786 cell) and humanized model
Identification of response biomarkers | Up to 24 months
  Characterization of the tumours using different techniques (RNASeq whole genome, NGS analysis, IHC, HTG focus RNAseq)
Identification of biomarkers of response | Evolution between inclusion and up to 24 months
  Immune status (Multi-IF analysis, TCR sequencing and clonality analysis, Anti-HERV T cell and humoral response)

CONTACTS AND LOCATIONS:
Overall Officials: BOYLE J Helen, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France